CLINICAL TRIAL: NCT00373815
Title: A Phase I Dose Escalation Study With Everolimus in Combination With Cyclosporine A and Prednisolone for the Treatment of Acute GVHD After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Everolimus in Combination With Cyclosporine A and Prednisolone for the Treatment of Graft Versus Host Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: high incidence of TTP, poor recrual
Sponsor: University Hospital Tuebingen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-002577-44
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Graft Versus Host Disease
Keywords: acute GVHD; Immunosuppression
MeSH Terms: conditions — Graft vs Host Disease | interventions — Everolimus

INTERVENTIONS:
Drug: Everolimus

SUMMARY:
The present protocol is a dose-finding and toxicity study in preparation of a randomised study comparing current standard treatment CSA/prednisolone with the new combination CSA/prednisolone/everolimus.

DETAILED DESCRIPTION:
The primary objective of the present study is to evaluate the feasibility of treatment with everolimus in combination with CSA/prednisolone in patients with aGVHD after allogeneic HSCT. This evaluation takes into account the following parameters:

* Feasibility of oral application everolimus
* Daily dose needed to reach the targeted plasma level everolimus
* Time to reach the targeted plasma level of everolimusSecondary objectivesThe study will evaluate the toxicity and safety of the treatment with ever-olimus/CSA/prednisolone with regard to
* Incidence and severity of treatment induced toxic events
* Incidence, severity and seriousness of adverse events
* Treatment induced morbidity
* Treatment induced 1-year-mortality Furthermore the study will collect data about
* Efficacy of everolimus/CSA/prednisolone on aGVHD
* Drug interactions between everolimus and CSA

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to inclusion into the study
* Allogeneic HSCT from HLA-identical related or unrelated donors
* Clinically confirmed acute GVHD ≥ grade II
* Age < 70 / > 18 years, male or female
* Karnofsky performance status > 60 %

Exclusion Criteria:

* Oral treatment is not feasible
* Severe hepatic impairment Child-Pugh C
* Active cerebral epilepsy
* Renal failure (Creatinine clearance < 50 ml/min)
* Life expectancy < 3 months
* Known hypersensitivity to everolimus, sirolimus or to any of the excipients
* Confirmed pregnancy (serum β-HCG)
* Non-effective contraception for both, male and female patients, if the risk of conception exists
* Patients with limited legal capacity
* Patients unwilling and unable to undergo study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-09; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of oral application everolimus
Daily dose needed to reach the targeted plasma level everolimus
Time to reach the targeted plasma level of everolimus

SECONDARY OUTCOMES:
Incidence and severity of treatment induced toxic events
Incidence, severity and seriousness of adverse events
Treatment induced morbidity
Treatment induced 1-year-mortality
Efficacy of everolimus/CSA/prednisolone on aGVHD
Drug interactions between everolimus and CSA

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang A Bethge, MD, Principal Investigator — Medical Center University of Tuebingen
Locations (1):
- Medical Center, Hematology & Oncology, University of Tuebingen, Tübingen, Germany

REFERENCES:
- See also: Related Info — http://www.onkologie-tuebingen.de